CLINICAL TRIAL: NCT06015906
Title: Guided Bone Regeneration Using Polydioxanone (PDO) Membrane in Sockets After Tooth Extraction: a Clinical Trial
Brief Title: Guided Bone Regeneration Using Polydioxanone (PDO) Membrane in Sockets After Tooth Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: M3 Health (Industry)
Collaborators: São Paulo State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Plenum Guide
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-10

CONDITIONS: Surgery, Oral
Keywords: Guided bone regeneration; Resorbable membrane; Plenum® Guide; Dental implant; Extraction socket preservation
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- socket (Sham Comparator): Tooth extraction socket filled only clot.
  Interventions: Procedure: Tooth extraction
- Socket associated with exposed absorbable membrane (Active Comparator): Socket filled with clot and covered with the Plenum® Guide membrane exposed in the intraoral region.
  Interventions: Device: Plenum® Guide; Procedure: Tooth extraction
- Socket associated with covered absorbable membrane (Active Comparator): Socket filled with clot and covered with the Plenum® Guide membrane and covered by mucosa (gingival tissue) in the intraoral region.
  Interventions: Device: Plenum® Guide; Procedure: Tooth extraction
- Socket filled with synthetic bone graft and covered absorbable membrane (Experimental): Socket filled with synthetic bone graft and the Plenum® Guide membrane covered by gingival tissue in the intraoral region.
  Interventions: Device: Plenum® Guide; Device: Plenum® Oss; Procedure: Tooth extraction
- Socket filled with synthetic bone graft and exposed absorbable membrane (Experimental): Socket filled with synthetic bone graft and Plenum® Guide membrane, where this membrane will be exposed in the intraoral region.
  Interventions: Device: Plenum® Guide; Device: Plenum® Oss; Procedure: Tooth extraction

INTERVENTIONS:
Device: Plenum® Guide — Plenum® Guide is a white, absorbable synthetic regenerative membrane composed of poly(dioxanone), which will be installed on the tooth extraction sockets.
  Other Names: PDO absorbable membrane
  Arms: Socket associated with covered absorbable membrane; Socket associated with exposed absorbable membrane; Socket filled with synthetic bone graft and covered absorbable membrane; Socket filled with synthetic bone graft and exposed absorbable membrane
Device: Plenum® Oss — Plenum® Oss is a synthetic bone graft based on biphasic calcium phosphate, which will be used to fill the tooth extraction sockets.
  Other Names: Synthetic bone graft
  Arms: Socket filled with synthetic bone graft and covered absorbable membrane; Socket filled with synthetic bone graft and exposed absorbable membrane
Procedure: Tooth extraction — Tooth extraction and subsequent surgical procedure of guided bone regeneration.
  Other Names: Guided bone regeneration

SUMMARY:
The goal of this clinical trial is to compare the maintenance of socket volume in the groups treated by a resorbable regenerative membrane (Plenum® Guide) covered or not with mucous tissue, with control without treatment. The main question it aims to answer is the effectiveness of the Plenum® Guide membrane in the process of guided bone regeneration, exposed or not, through the preservation and neoformation of bone tissue in the tooth extraction socket procedures.

DETAILED DESCRIPTION:
Patients will be submitted to tooth extraction, the surgical procedure of guided bone regeneration using regenerative membranes and synthetic bone graft, and subsequent installation of dental implants. The 05 groups will be compared to observe if the proposed medical devices effectively will maintain the socket's bone volume during the healing phase before the installation of the dental implants (1. socket filled only with clot, 2. socket associated with exposed absorbable membrane, 3. socket associated with covered absorbable membrane, 4. socket filled with synthetic bone graft and covered absorbable membrane, 5. socket filled with synthetic bone graft and exposed absorbable membrane).

ELIGIBILITY:
Inclusion Criteria:

* Possess the four bone walls after the extraction procedure;
* Over 18 years old;
* And who have signed the TCLE.

Exclusion Criteria:

* Uncontrolled systemic impairments;
* Teeth in areas of tumor lesions;
* Acute infectious processes;
* Deciduous dental elements;
* Untreated periodontal problems;
* Smokers;
* Radiated in the head or neck region;
* Allergy to any component used in the research;
* Psychological disorders;
* Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Rate of alveolar repair | Comparison of exams obtained in the preoperative period, immediate postoperative period (7 days) and late postoperative period (3 months)
  Accessed via cone beam computed tomography
Rate of newly formed bone tissue, soft tissue and residual bone graft material | 4 months after extraction
  immunohistochemical analyzes of histological sections

CONTACTS AND LOCATIONS:
Overall Officials: Sybele Saska Specian, PhD, Study Director — Study Director

IPD SHARING:
Plan to Share IPD: No